CLINICAL TRIAL: NCT04438681
Title: INSTIGO Trial: Evaluation of a Plasma Protein Profile as a Predictive Biomarker for Metastatic Relapse in Triple Negative Breast Cancer Patients
Brief Title: Evaluation of a Plasma Protein Profile as a Predictive Biomarker for Metastatic Relapse in Triple Negative Breast Cancer Patients
Acronym: INSTIGO
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01423-36
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The INSTIGO study aims to assess a plasma protein profile at different stages of patient follow-up as a predictive factor of metastatic recurrence in triple negative breast cancer. It also aims to look at other potential biomarkers of metastatic relapse such as Tumor-infiltrating Lymphocytes, circulating tumor DNA, figurative elements in blood, or a tumor RNA signature.

DETAILED DESCRIPTION:
The investigators propose to carry out a study that measures the concentrations of a set of plasma proteins in order to assess their ability to predict metastatic relapse of triple negative breast cancer. A plasma protein profile could be an interesting biomarker since it is easily accessible and quantifiable.

The investigators also propose to search relation between metastatic relapse in TNBC and other biomarkers or potential biomarkers such as Tumor-infiltrating Lymphocytes (TILs), figurative blood components and circulating tumour DNA (ctDNA).

Finally, they also want to validate a TNBC RNA signature, established at Jean PERRIN Center, by analyzing the RNA expression of 8 genes.

Before treatment begins, the patient will take an initial blood sample. A second blood sample will be taken on the day of the first surgery or the day of the surgery post chemotherapy. A third blood sample will be done on the day of the beginning of the radiotherapy. A 4th and a 5th blood sample will be done at 6 months and 1 year respectively after the end of the radiotherapy. A part of these blood samples will be used for the quantification of circulating proteins, for the determination of the blood's figurative elements and for the quantification of circulating tumour DNA.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18 years
* Diagnosed with primitive, non-metastatic, histologically proved, triple negative breast cancer
* Patient able to understand the French language
* Patient affiliated to social security
* Obtaining signed written consent

Exclusion Criteria:

* Persons deprived of their freedom or under guardianship or incapable of giving consent
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with primitive, non-metastatic, histologically proved, triple negative breast cancer
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2026-11-09 (Estimated); Study Completion 2029-11-09 (Estimated)

PRIMARY OUTCOMES:
Identification at diagnosis of a plasma protein profile predictive of metastatic relapse in patients with triple-negative breast cancer (TNBC) | 8 years
  - Plasma concentrations of a set of proteins at diagnosis (measured in g/L)
Identification at diagnosis of a plasma protein profile predictive of metastatic relapse in patients with triple-negative breast cancer (TNBC) | 8 years
  - Time to metastatic relapse

SECONDARY OUTCOMES:
Identification of a plasma protein profile predictive of metastatic relapse in patients with TNBC : on the day of primary surgery or post-chemotherapy surgery, the day the radiotherapy begins, at 6 months after radiotherapy and one year post-radiotherapy | 8 years
  - Plasma concentrations of a set of proteins (measured in g/L)
Identification of a plasma protein profile predictive of metastatic relapse in patients with TNBC : on the day of primary surgery or post-chemotherapy surgery, the day the radiotherapy begins, at 6 months after radiotherapy and one year post-radiotherapy | 8 years
  - Time to metastatic relapse
Identification of a characteristic plasma protein profile at the time of metastatic relapse | 8 years
  - Plasma concentrations of a set of proteins (measured in g/L)
Evaluation of the relationship between the rate of tumour lymphocyte infiltration at diagnosis and metastatic relapse. | 8 years
  - Tumor lymphocyte infiltration rate before treatment
Evaluation of the relationship between ctDNA plasma levels and metastatic disease relapse | 8 years
  - Measurement of plasma ctDNA level
Evaluation of the relationship between ctDNA plasma levels and metastatic disease relapse | 8 years
  - Time to metastatic relapse
Evaluation of the relationship between Platelet-to-lymphocyte Ratio (PLR) and Neutrophil-to-lymphocyte Ratio (NLR) and metastatic relapse | 8 years
  - The values of NLR and PLR at diagnosis (no Unit)
Evaluation of a metastatic relapse prognostic RNA signature for triple negative breast tumors | 8 years
  - RNA expression of 6 genes of interest
Identification at diagnosis of a plasma protein profile predictive of response to neoadjuvant chemotherapy | 3 years and 6 months
  - Plasma concentrations of a set of proteins at diagnosis
Identification at diagnosis of a plasma protein profile predictive of response to neoadjuvant chemotherapy | 3 years and 6 months
  - Histological response according to the Sataloff classification
Evaluation of the relationship between the rate of tumour lymphocyte infiltration at diagnosis and the response to a neoadjuvant chemotherapy . | 3 years and 6 months
  - Tumor lymphocyte infiltration rate before treatment
Evaluation of the relationship between Platelet-to-lymphocyte Ratio (PLR) and Neutrophil-to-lymphocyte Ratio (NLR) and the response to a neoadjuvant chemotherapy | 3 years and 6 months
  * The values of NLR and PLR at diagnosis
  * The values of NLR and PLR after neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Jean PERRIN, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pinard C, Ginzac A, Molnar I, Veyssiere H, Bidet Y, Sapin V, Durif J, Abrial C, Penault-Llorca F, Durando X, Radosevic-Robin N. Identification of serum proteins associated with response of triple-negative breast cancer to neoadjuvant chemotherapy: preliminary results from the INSTIGO trial. Clin Proteomics. 2025 Dec 29;22(1):50. doi: 10.1186/s12014-025-09574-0. PMID 41462069
- [Derived] Veyssiere H, Lusho S, Molnar I, Kossai M, Bernadach M, Abrial C, Bidet Y, Radosevic-Robin N, Durando X. INSTIGO Trial: Evaluation of a Plasma Protein Profile as a Predictive Biomarker for Metastatic Relapse of Triple Negative Breast Cancer. Front Oncol. 2021 Jun 25;11:653370. doi: 10.3389/fonc.2021.653370. eCollection 2021. PMID 34249690